CLINICAL TRIAL: NCT00005435
Title: Hostility and Pathogenic Mechanisms of Coronary Heart Disease in Women
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4362; R29HL046283 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To determine the combined effects of hostility, harassment, lipids, and oral contraceptive (0C) use on physiological responses in young and middle-aged premenopausal women.

DETAILED DESCRIPTION:
BACKGROUND:

Preliminary findings already have shown that, in contrast to women with low scores on the Cook and Medley Hostility (Ho) scale, women with high Ho scores exhibit greater cardiovascular changes to harassment. Additional findings have suggested that oral contraceptive (0C) use may also be associated with increased behaviorally-induced physiological changes, especially in low Ho women. Similarly, higher levels of total serum cholesterol (TSC) have been positively associated with greater stress-induced neurohormonal changes in middle-aged men with high Ho scores.

DESIGN NARRATIVE:

Assessment of autonomic activity took place in the laboratory and during a 24 hour ambulatory measurement period. Hostility was measured with the Cook and Medley Hostility scale. The laboratory assessment helped to determine if high hostility women responded to harassment with greater cardiovascular and neurohormonal changes than low hostility women, and if this relationship was altered by 0C use, lipids, and age. The ambulatory assessment of autonomic activity allowed an exploration of the responses of high and low hostility subjects to daily-life stressors. Several hypothesis were explored: 1) Did harassment produce neuroendocrine as well as cardiovascular hyperreactivity in young women, and did this hyperreactivity generalize from laboratory to real-life? 2) Were the harassment-induced cardiovascular and neuroendocrine changes in young women also present in middle-aged women? 3) To what extent did 0C use modulate the cardiovascular and neuroendocrine responses to harassment in young women, and was 0C use also altering the hostility--related associations between lipids and reactivity? 4) Were the differential lipid-reactivity associations observed in middle-aged men as a function of high and low hostility scores present in women, and, if so, were they modulated by age?

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-07; Study Completion 1997-06 (Actual)

REFERENCES:
- [Background] Harralson TL, Suarez EC, Lawler KA. Cardiovascular reactivity among hostile men and women: the effects of sex and anger suppression. Womens Health. 1997 Summer;3(2):151-64. PMID 9332156
- [Background] Suarez EC, Harlan E, Peoples MC, Williams RB Jr. Cardiovascular and emotional responses in women: the role of hostility and harassment. Health Psychol. 1993 Nov;12(6):459-68. doi: 10.1037//0278-6133.12.6.459. PMID 8293729
- [Background] Suarez EC. Relations of trait depression and anxiety to low lipid and lipoprotein concentrations in healthy young adult women. Psychosom Med. 1999 May-Jun;61(3):273-9. doi: 10.1097/00006842-199905000-00004. PMID 10367605
- [Background] Suarez EC, Bates MP, Harralson TL. The relation of hostility to lipids and lipoproteins in women: evidence for the role of antagonistic hostility. Ann Behav Med. 1998 Spring;20(2):59-63. doi: 10.1007/BF02884449. PMID 9989309